CLINICAL TRIAL: NCT02245126
Title: The Use of Lignocaine and Bupivacaine Mix in Adult Safe Male Circumcision; Less is More
Brief Title: The Use of Lignocaine and Bupivacaine Mix in Adult Safe Male Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hospital Kampala (Other)
Collaborators: Makerere University (Other)
Responsible Party: Principal Investigator, Moses Galukande, director of Surgery, International Hospital Kampala
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC REF 2014-050
Record Dates: First submitted 2014-08-02; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Post Operative Pain
Keywords: Pain, Visual analogue scale
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lignocaine-bupivacaine lower dosage mix (Experimental): Men who received the 3-3-4 local anaesthetic mix( 3 cc of lignocaine 2% , 3cc of bupivacaine 0.5% and 4cc of water for injection)
  3-3-4 mix was administered
  Interventions: Drug: 3-3-4 mix
- Lignocaine-bupivacaine higher dosage mix (Active Comparator): In this group (4-4-2 group) eligible men were receiving an injection of the 4-4-2 local anesthetic mix ( composed of 4cc of parental lignocaine 2%, 4cc of parental bupivacaine 0.5% and 2cc of water for injection). This mix is given once before commencement of the surgical procedure safe male circumcision.
  Interventions: Drug: 4-4-2

INTERVENTIONS:
Drug: 3-3-4 mix — the drug mix included lidocaine, bupivacaine and water for injection
  Other Names: Lidocaine; Bupivaciane
  Arms: Lignocaine-bupivacaine lower dosage mix
Drug: 4-4-2 — In this group (4-4-2 group) eligible men were receiving an injection of the 4-4-2 local anesthetic mix ( composed of 4cc of parental lignocaine 2%, 4cc of parental bupivacaine 0.5% and 2cc of water for injection). This mix is given once before commencement of the surgical procedure safe male circumcision.
  Other Names: Lidocaine; Bupivacaine
  Arms: Lignocaine-bupivacaine higher dosage mix

SUMMARY:
Using routinely collected data to compare different concentrations of locally applied anaesthetic drugs and determine which concentrations give better pain control during voluntary medical Male circumcision.

DETAILED DESCRIPTION:
The objective of this study therefore was to assess self-reported pain and adverse events when using two different concentrations of lignocaine and bupivacaine mixture while performing routine safe medical circumcision (SMC).

Methods Design This was an observational analytical study.

Setting At an urban high volume SMC site in a resource limited setting, over a 6 weeks period.

Participants Adult males aged18 - 49 years presenting for routine voluntary SMC were recruited for enrollment. All men were offered voluntary HIV counseling and testing before the surgery, received group counseling /health education on HIV prevention, were offered HIV testing, individual counseling where necessary to address questions and to clarify any queries, and free condoms were available. All participants were screened for contraindications to SMC such as active sexual transmitted infections (STI), commonly manifesting as urethral discharge or penile ulcers.

Ethical consideration All participants after they were counselled and provided written informed consent. Ethical approval was obtained from the Makerere College of Health Sciences Ethics and Research Committee.

Lignocaine and Bupivacaine (LiB) mixtures and procedure Lignocaine 2% and bupivacaine 0.5% were procured locally, from suppliers licensed and approved by the national drug authority (NDA), and was within the expiry date. The 4-4-2 mix was 4cc of Lignocaine 2%, 4cc of 0.5% bupivacaine and 2cc of water for injection, all drawn into a 10cc syringe. The 3-3-4 mix was 3cc of Lignocaine 2%, 3cc of bupivacaine 0.5% and 4 cc of water for injection.

We assigned participants to the two groups (each group on alternative weeks). We administered additional local analgesia for those who experienced break-through pain during the procedure. We recorded the mix ratio, the time the procedure commenced and ended using a stop clock, presence of break-through pain during SMC, and pain at 30 and 60 minutes after SMC (post-operative). We encouraged clients to report pain and a visual analogue score (VAS) pain chart was used to estimate pain intensity. Post-operative pain was graded as mild if the VAS score were 0-5, moderate if scores were 6-8 and severe if 9-10. We monitored the clients in the recovery room for additional post-operative pain and oral analgesia were given when and if was needed.

Other adverse events: participants were observed for central nervous system (CNS) toxicity, convulsions, coma and respiratory depression and cardiovascular system (CVS) toxicity Bradycardia pulse rate < 60bpm (beats per minute)

ELIGIBILITY:
Inclusion Criteria:

* all adult male aged18 and 49 years

Exclusion Criteria:

* severe comorbid states such as sickle cell disease
* uncontrolled diabetes
* hypertension
* active sexually transmitted infections and genital ulcers
* in addition known allergy to lidocaine or bupivacaine

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
pain score | immediate post operative period
  measure at intervals after the procedure is completed

CONTACTS AND LOCATIONS:
Overall Officials: Moses Galukande, MD, Principal Investigator — International Hospital
Locations (1):
- International Hospital Kampala, Kampala, Kampala, Uganda

REFERENCES:
- [Derived] Galukande M, Nakaggwa F, Busisa E, Sekavuga Bbaale D, Nagaddya T, Coutinho A. Long term post PrePex male circumcision outcomes in an urban population in Uganda: a cohort study. BMC Res Notes. 2017 Oct 30;10(1):522. doi: 10.1186/s13104-017-2845-9. PMID 29084559